CLINICAL TRIAL: NCT07317986
Title: CommuniT1D: A Customized Virtual Peer Support Program For People Living With Type 1 Diabetes In Canada
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CommuniT1D
Record Dates: First submitted 2025-12-19; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-09

CONDITIONS: Type 1 Diabetes (T1D)
Keywords: peer support
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CommuniT1D arm (Experimental): People in the intervention will be offered a peer support intervention consisting of monthly Zoom meetings with peers in similar situations.
  Interventions: Other: Peer support meetings

INTERVENTIONS:
Other: Peer support meetings — Online videoconference meetings held approximately monthly.

SUMMARY:
When you live with type 1 diabetes (T1D), it is easy to feel alone. Managing your own T1D or your child's T1D takes constant effort that is invisible to most people. Often, the only people who really understand what you are going through are other people in similar situations, but it's hard to find those people, especially when there are other aspects of your life that might be different from others with T1D. For example, you might have a very young child with T1D, you might be racialized and deal with racism in health care on top of T1D, you might be going through menopause with T1D, you might be aging out of provincial or parental device coverage, you might speak a different language from most people around you with T1D, or any one of many other things that make your situation unique. This project aims to create regular, small online meetings via Zoom or similar technologies to bring together people across Canada who are managing T1D (their own and/or their child's) who have other things in common. We will create these small groups that will meet monthly as well as larger monthly webinars covering topics of interest. We will track how people like the groups, how they feel, what they like and don't like, and adjust the program accordingly. This project is led by researchers and others who themselves live with T1D. We believe that this kind of peer support can be extremely helpful to people with T1D and it will provide needed mental health support.

DETAILED DESCRIPTION:
Background and objectives: Type 1 diabetes (T1D) is a largely self-managed condition that requires ongoing daily tasks and decisions. Many people living with T1D in Canada manage it alone, which can feel very isolating and negatively affect physical and mental health. Connecting with other people in similar situations may help to reduce the potential burden associated with managing this health condition. We aim to co-develop and evaluate a virtual peer support program called CommuniT1D, led by people with T1D, to improve the overall wellbeing of people across Canada whose lives are affected by T1D.

Methods and analysis: Using a community-based participatory design and action research approach and a realist evaluation framework, we will first co-develop CommuniT1D by working together as a group of people with T1D, researchers, and clinicians. Over two thirds of steering committee members live with T1D (their own or their child's.) This collective lived expertise is complemented by experts in mental health, social support, health services research, and other relevant fields. Once the program is ready to welcome members, we will work with our partner organizations, networks, and use tailored ads to recruit CommuniT1D peer leaders and members. We will then form virtual peer support groups of people with shared lived experience. Within the program, we will hold monthly small group meetings led by peer leaders via an online platform. We will also hold monthly large webinars open to all CommuniT1D members and other interested people. To evaluate CommuniT1D, we will conduct surveys at baseline and every 6 months, collecting data about diabetes distress, life challenges, quality of life, wellbeing, management indicators, and access and use of management tools and services. We will analyze quantitative data using repeated measures analysis of variance. We will also conduct individual interviews with CommuniT1D members and peer leaders at two time points. We will analyze interview data thematically, and create a logic model by triangulating results from qualitative and quantitative analyses, applying a realist evaluation lens.

Discussion: Peer support may help people with T1D feel less alone and better supported. This protocol outlines the design of a virtual peer support program called CommuniT1D to improve the wellbeing of people whose lives are affected by T1D in Canada. We hope that this program will help better equip people with T1D to cope with T1D-related stressors, thus improving the lives of people with T1D in Canada.

ELIGIBILITY:
Inclusion Criteria: Participants in CommuniT1D must be people living with T1D or another rare, insulin-requiring form of diabetes, namely, Latent autoimmune diabetes of adults (LADA), Maturity-Onset Diabetes of the Youth (MODY), or type 3c, which occurs due to an injury to or removal of the pancreas. Loved ones such as a parent, child, spouse, caregiver, or friend of an individual with T1D or other rarer forms of diabetes will also be eligible to participate in CommuniT1D. Participants must be 18 years and older, reside in Canada, and be able to read the consent form in English or French.

Exclusion Criteria: Individuals with type 2 diabetes, pre-diabetes, or gestational diabetes and no connection to T1D, LADA, MODY, type 3c, or other rare, insulin-requiring forms of diabetes will not be included in CommuniT1D. Individuals under 18 years old will also be ineligible to participate. As the program grows, we hope to expand to also include adolescents and children, who may need parental consent for them to join, depending on their Canadian province or territory of residence. Should we be able to pursue this option, we will work with institutional research ethics boards to ensure that we welcome participation by youth while also ensuring their safety within CommuniT1D. In such a case, the age restrictions in our eligibility criteria would change.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-07-07 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
Diabetes Distress | Every 6 months from enrollment to the end of intervention (estimated 2 years)
  We will use the Type 1 Diabetes Distress Scale [PMID: 25765489] and work with our steering committee to adapt the scale in order to address specific life situations relevant to our participants. For example, for CommuniT1D members who are employed, we will add two additional questions about work-related diabetes distress. [PMID: 29604390] For parents of teens with T1D, we will use the Parent Diabetes Distress Scale (PARENT-DSS) [https://behavioraldiabetes.org/scales-and-measures/#1448434808823-e055c4f8-b047] and will adapt this scale for parents of younger children with T1D. For partners of individuals with T1D, we will use the Partner Diabetes Distress Scale (PARTNER-DDS). [https://behavioraldiabetes.org/scales-and-measures/#1448434936830-83758e0b-2ee4] Lower diabetes distress scores are considered desirable compared to higher scores.

SECONDARY OUTCOMES:
Caregiver Stress | Every 6 months from enrollment to the end of intervention (estimated 2 years)
  For participants who identify as caregivers of a person living with T1D, we will use the Kingston Caregiver Stress Scale. [http://www. kingstonscales.org/caregiver-stress-scale.htm]
Anxiety and Depression | Every 6 months from enrollment to the end of intervention (estimated 2 years)
  We will measure symptoms of anxiety and depression using the Hospital Anxiety and Depression Scale (HADS). [PMID: 6880820]
Self-Efficacy | Every 6 months from enrollment to the end of intervention (estimated 2 years)
  We will evaluate diabetes-specific self-efficacy using the Confidence in Diabetes Scale, which measures participants' confidence in their ability to perform essential diabetes self-care activities. [PMID: 12610027]
Fear of Hypoglycemia | Every 6 months from enrollment to the end of intervention (estimated 2 years)
  To examine fear of hypoglycemia, we will use the short form of the Hypoglycemia Fear Survey II, a validated tool that captures behavioral and emotional responses related to hypoglycemic episodes. [PMID: 27278467]
Well-Being | Every 6 months from enrollment to the end of intervention (estimated 2 years)
  We will assess general psychological well-being with the WHO-5 Well-Being Index. This brief instrument has demonstrated high sensitivity for detecting depressive symptoms and is validated in populations with T1D. [PMID: 17475940]
Diabetes-Specific Quality of Life | Every 6 months from enrollment to the end of intervention (estimated 2 years)
  We will measure diabetes-specific quality of life using the Audit of Diabetes-Dependent Quality of Life (ADDQoL). [PMID: 10457741]
Perceived Social Support | Every 6 months from enrollment to the end of intervention (estimated 2 years)
  To capture perceived social support, we will use a 5-item adaptation of the Social Provisions Scale developed specifically for Canadian populations. [https://doi.org/10.24095/hpcdp.39.12.02]
Self-Compassion | Every 6 months from enrollment to the end of intervention (estimated 2 years)
  We will measure self-compassion using the Self-Compassion Scale-Short Form (SCS-SF). [https://doi.org/10.1080/15298860309027]

OTHER OUTCOMES:
Unmet Needs for Care | Every 6 months from enrollment to the end of intervention (estimated 2 years)
  To assess unmet needs for care, we will use selected items adapted from the Canadian Community Health Survey (CCHS). [https://www23.statcan.gc.ca/imdb/p2SV.pl?Function=getSurvey&SDDS=3226] These items will allow us to identify perceived gaps in access to appropriate and timely diabetes-related care.
Personality Traits | Every 6 months from enrollment to the end of intervention (estimated 2 years)
  We will use the Ten-Item Personality Inventory (TIPI) to describe participants' personality traits. [https://doi.org/10.1016/S0092-6566(03)00046-1] While not a direct outcome measure, this tool will allow us to explore how individual personality profiles may moderate the effects of the intervention, and may also capture shifts in constructs such as conscientiousness, which may be useful for diabetes management.

CONTACTS AND LOCATIONS:
Locations (1):
- Université Laval, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data will be shared on Borealis (Université Laval's Dataverse instance.)
Supporting Information: Study Protocol, ICF
Time Frame: After the study is complete.
Access Criteria: Anyone with Internet access will be able to access all public-facing information.
URL: https://borealisdata.ca/dataverse/laval